CLINICAL TRIAL: NCT01264484
Title: ADVANTAGE Prosthetic Heart Valve Long Term Follow Up
Brief Title: ADVANTAGE® Prosthetic Heart Valve Long-term Follow-up Trial
Status: Terminated | Type: Observational
Why Stopped: The primary objective was considered sufficient for follow-up.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: ADVANTAGE
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Heart Valve Stenosis
Keywords: Advantage; Non-interventional; Post market release study; Germany; Treated with Advantage prosthetic heart valve

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advantage prosthetic heart valve: All patients who were enrolled and implanted with an Advantage valve in the Herzzentrum Nordrhein-Westfalen (Bad Oeynhausen, Germany) and Deutsches Herzzentrum München (Munich, Germany) during the previous Advantage clinical study study and who agree to participate in this long-term follow-up study by informed consent.
  Interventions: Device: Advantage Prosthetic Heart Valve

INTERVENTIONS:
Device: Advantage Prosthetic Heart Valve — All patients eligible for this study are treated with an Advantage prosthetic heart valve

SUMMARY:
The objective of this study is to assess long term safety and durability of the Advantage prosthetic heart valve.

DETAILED DESCRIPTION:
The objective of this study is to assess long term safety and durability of the Advantage prosthetic heart valve in patients who were already implanted with this device.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the ADVANTAGE Prosthetic Heart Valve Study in Herz- und Diabeteszentrum (Bad Oeynhausen) or Deutsches Herzzentrum (Munich)
* Signed and dated patient data release form
* Available for follow-up

Exclusion Criteria:

* High probability of non-adherence to physician's follow-up requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population for this study includes all patients who were already enrolled in the ADVANTAGE Prosthetic Heart Valve Study in two German Centers and are still available for follow-up
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Long-term safety and durability of the valve | 5 year follw-up
  The long-term safety of the valve will be assessed by the rate of valve related complications. The long-term durability of the valve will be assessed by measuring hemodynamic performance of the valve

CONTACTS AND LOCATIONS:
Overall Officials: Rudiger Lange, Prof. Dr., Principal Investigator — Deutsches Herzzentrum München; Jan Gummert, prof. dr., Principal Investigator — Herzzentrum Nordrhein-Westfalen, Bad Oeynhausen
Locations (2):
- Germany (2):
  - Herz- und Diabetescentrum Bad Oeynhausen, Bad Oeynhausen
  - Deutsches Herzzentrum Munchen, München

REFERENCES:
- See also: general Medtronic website — http://www.medtronic.com